CLINICAL TRIAL: NCT02692742
Title: A Randomised, Double-Blind, Placebo-Controlled, Parallel-Design, Multi-Center Study to Investigate the Efficacy To Reduce Chemotherapy-Induced Neutropenia (CIN), Effects on the Haematopoietic System, Safety and Pharmacokinetics of Myelo001 in Patients Receiving Adjuvant or Neoadjuvant Chemotherapy for the Treatment Of Breast Cancer
Brief Title: Efficacy and Safety Phase IIa Study of Myelo001 in Chemotherapy-Induced Neutropenia
Acronym: MyeloConcept
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Myelo Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CT-MT001-2-2015-1; 2015-003610-25 (EudraCT Number)
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Chemotherapy-Induced Neutropenia; Myelosuppression; Breast Cancer
Keywords: Chemotherapy; Chemotherapy-induced Neutropenia; Supportive Care; Myelosuppression; CIN
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Myelo001 (Experimental): Myelo001 100 mg QD
  Interventions: Drug: Myelo001
- Placebo (Placebo Comparator): Matching Placebo QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Myelo001 — Intake of study drug once daily per os for a maximum of 28 days in addition to Epirubicin and Cyclophosphamide treatment
  Arms: Myelo001
Drug: Placebo — Intake of study drug once daily per os for a maximum of 28 days in addition to Epirubicin and Cyclophosphamide treatment
  Arms: Placebo

SUMMARY:
Neutropenia is the most serious hematologic toxicity of cancer chemotherapy, often limiting the doses and density of chemotherapy that can be tolerated. The degree and duration of neutropenia determine the risk of infection. Myelo001, a small orally bioavailable molecule, has been shown in chemotherapy- or radiotherapy-induced myelosuppression to stimulate differentiation of peripheral white blood cells (WBC) and bone marrow cells of the leucocytic, lymphocytic, and erythrocytic lineage. The purpose of the MyeloConcept study is to determine the safety and effectiveness of Myelo001 in preventing or reducing chemotherapy-induced neutropenia and myelosuppression in patients receiving chemotherapy due to breast cancer.

DETAILED DESCRIPTION:
Phase IIa study, 1:1 randomized, double-blind, placebo-controlled, parallel-design, multi-center study. Each breast cancer patient will be randomly assigned into one of two treatment arms receiving either Myelo001 or placebo as a tablet. Investigational medicinal product is taken as supportive care for 23 consecutive days during chemotherapy treatment. Hematologic and safety parameters as well as actual begin and doses of following chemotherapy cycles will be assessed. A single primary variable will be analyzed with test statistics based on frequent absolute neutrophil measurements. Additionally, in a subgroup of patients biomarkers and pharmacokinetics of Myelo001 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient of any racial origin having fulfilled her 18th birthday on Visit 1 (Screening)
2. Histologically confirmed invasive breast cancer scheduled for neoadjuvant or adjuvant chemotherapy (patient with primary wound healing ([R0])
3. Already selected for neoadjuvant or adjuvant standard of care EC regimen (Epirubicin 90 mg/m2 BSA (body surface area) + Cyclophosphamide 600 mg/m2 BSA q21d (every 21 days)) (with or without treatment with taxanes afterwards)
4. Risk of chemotherapy-induced Febrile Neutropenia ≤20% according to ASCO Guidelines (2015)
5. More than 5 days remaining before the planned initiation of the 1st chemotherapy cycle
6. Performance status Grade 0-1 (ECOG)
7. Echocardiography: No contraindication for the scheduled chemotherapy
8. Haematologic, laboratory and chemistry thresholds at baseline:

   * Absolute neutrophil count (ANC) ≥2,000 cells/ mm3 (≥2.0 x 10/L)
   * Platelet count ≥100,000/mm3 (≥100 x 10exp9/L)
   * Haemoglobin ≥10 g/dL
   * Total bilirubin <1.5 x, AST, ALT <2.5 x upper limit of normal (ULN)
   * Serum creatinine <2.0 mg/dL
9. Able to read, understand and willing to sign the informed consent form
10. Able to undergo the investigations and to follow the Visit schedule

Exclusion Criteria:

1. Suspected allergy to Myelo001 or its excipients
2. Prior chemotherapy
3. Prior or concomitant treatment with radiotherapy
4. Currently on or scheduled for other immunomodulatory or immunosuppressive therapies (e.g. TNF inhibitors) during the first chemotherapy cycle
5. Currently on or scheduled for other immunostimulatory or hematopoietic active therapies (e.g.G-CSF, GM-CSF)
6. Currently on or scheduled for primary prophylaxis with antibiotics in the first chemotherapy cycle
7. History of bone marrow transplantation or stem cell transplant
8. Administration of another investigational medicinal product / medical device within 30 days prior to screening. Participation in non-interventional, national or international cancer registries is allowed.
9. Already confirmed HIV, hepatitis B or C virus (HBV or HCV) infection
10. History of somatic disease/condition that may interfere with the objectives of the study
11. Any other medical disease or clinical laboratory parameter outside the normal range and of clinical significance according to the investigator
12. Serious uncontrolled comorbidities
13. Pregnant or breast-feeding subject
14. Woman considered to be of childbearing potential who do not use highly effective birth control methods during the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Threshold area over the curve (AOC1) of ANC: Area below the threshold line (ANC 2.0x10^9/L classified as grade 1 neutropenia) and above the individual ANC trajectory | visit 3 to visit 10 (22 days)
Threshold area over the curve (AOC3) of ANC: Area below the threshold line (ANC 1.0x10^9/L classified as grade 3 neutropenia) and above the individual ANC trajectory | visit 3 to visit 10 (22 days)
Duration of ANC < 1.0x10^9/L classified as grade 3 neutropenia | visit 3 to visit 10 (22 days)

SECONDARY OUTCOMES:
Treatment success rate: a) Neutropenia grade ≤2, b) No need for G-CSF rescue therapy, c) No early withdrawal (drop-out). | visit 3 to visit 10 (22 days)
Threshold AOC of ANC (AOC4): Area below the threshold line (ANC 0.5x10^9/L classified as grade 4 neutropenia) and above the individual ANC trajectory | visit 3 to visit 10 (22 days)
Change of Threshold Area over the Curve of lymphocytes | visit 3 to visit 10 (22 days)
Change of Threshold Area over the Curve of leukocytes | visit 3 to visit 10 (22 days)
Change of Threshold Area over the Curve of thrombocytes | visit 3 to visit 10 (22 days)
Proportion of patients with neutropenia grade 1 and higher; 3 and higher, 4, and ANC ≤0.1x 10^9/L | visit 3 to visit 10 (22 days)
Duration of neutropenia grade 1 and higher; 3 and higher, 4, and ANC ≤0.1x 10^9/L | visit 3 to visit 10 (22 days)
ANC at nadir | visit 3 to visit 10 (22 days)
Time to ANC nadir (from start of chemotherapy) | visit 3 to visit 10 (22 days)
Time to ANC recovery from grade 3 neutropenia, i. e. time from onset to time of reaching neutropenia grade ≤2 (ANC ≥ 1.5x10^9/L) | visit 3 to visit 10 (22 days)
Time to ANC recovery from grade 4 neutropenia, i. e. time from onset to time of reaching neutropenia grade ≤2 (ANC ≥ 1.5x10^9/L) | visit 3 to visit 10 (22 days)
Time to ANC recovery from profound neutropenia (ANC ≥ 0.1x10^9/L), i. e. time from onset to time of reaching neutropenia grade ≤2 (ANC ≥1.5x10^9/L) | visit 3 to visit 10 (22 days)
Proportion of patients with rescue therapy | visit 3 to visit 10 (22 days)
Proportion of patients developing febrile neutropenia (body temperature ≥38.3°C by single tympanic or oral measurement) and ANC ≤0.5x 10^9/L (Grade 4) | visit 3 to visit 10 (22 days)
Proportion of patients with CTX dose reduction and/or delay of CTX cycle 2 | visit 10 to visit 11

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Pleimes, MD, Study Director — Myelo Therapeutics GmbH
Locations (23):
- Germany (23):
  - Site 20, Aachen
  - Site 16, Aurich
  - Site 21, Dresden
  - Site 26, Dresden
  - Site 05, Erlangen
  - Site 09, Esslingen am Neckar
  - Site 02, Frankfurt a.M.
  - Site 13, Frankfurt a.M.
  - Site 01, Friedrichshafen
  - Site 25, Goslar
  - Site 11, Hamburg
  - Site 10, Hanover
  - Site 22, Hanover
  - Site 07, Konstanz
  - Site 29, Lübeck
  - Site 03, Mainz
  - Site 23, Mainz
  - Site 04, Offenbach
  - Site 19, Oldenburg
  - Site 17, Ravensburg
  - Site 24, Rosenheim
  - Site 28, Tübingen
  - Site 12, Westerstede

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company homepage — http://www.myelotherapeutics.com